CLINICAL TRIAL: NCT02826902
Title: Effect of Anesthesia on Quality of Recovery in Patients Undergoing Correctional Tibial Osteotomy - A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 4-2016-0164
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Short Stature; Osteoarthritis
Keywords: Total intravenous anesthesia; desflurane; QoR-40; correctional tibial osteotomy
MeSH Terms: conditions — Dwarfism; Osteoarthritis | interventions — Propofol; Remifentanil; Desflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TIVA group (Active Comparator)
  Interventions: Drug: propofol and remifentanil
- Inhalation anesthesia group (Active Comparator)
  Interventions: Drug: desflurane and remifentanil

INTERVENTIONS:
Drug: propofol and remifentanil — Anesthesia is induced and maintained by effect-site target controlled infusion of propofol and remifentanil
  Arms: TIVA group
Drug: desflurane and remifentanil — Anesthesia is induced and maintained with desflurane and remifentanil
  Arms: Inhalation anesthesia group

SUMMARY:
The effect of total intravenous anesthesia (TIVA) versus inhalational anesthesia on the quality of recovery from surgery has been reported in several different types of operations. The Quality of Recovery 40 (QoR-40) questionnaire is designed multi-dimensionally to assess the degree of recovery after anesthesia and surgery, and has been validated in previous studies. The present study aims to compare the quality of recovery with the QoR-40 questionnaire, in patients undergoing correctional tibial osteotomy under general anesthesia with either TIVA with propofol or inhalational anesthesia with desflurane.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients over the age of 19 scheduled for cosmetic lower limg lengthening for short stature, or correctional tibial osteotomy for osteoarthritis

Exclusion Criteria:

1. Patient refusal
2. Patients with altered mental status
3. Ejection fraction under 55%
4. Recent MI, CVA, or major cardiovascular surgery
5. 3rd degree AV block, 2nd degree AV block with P:QRS ration greater than 3:1
6. Hemodynamically unstable patients requiring vasopressors or oxygen therapy
7. Febrile patients
8. Patients with decreased renal function (serum Cr > 0.1 mg/dL)
9. Patients with known allergies to propofol
10. Pregnant patients

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2019-11-09 (Actual); Study Completion 2019-11-09 (Actual)

PRIMARY OUTCOMES:
QoR-40 score | 24 hours after surgery

SECONDARY OUTCOMES:
QoR-40 score | preoperative period to 48 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No